CLINICAL TRIAL: NCT01133392
Title: Evaluation of the Bioequivalence of Two Formulations of Insulin Lispro in Healthy Subjects
Brief Title: Bioequivalence of Two Lispro Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13300; F3Z-EW-IOPY (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Volunteers
Keywords: insulin; lispro
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro A (Experimental): 20 units (U) subcutaneously (SC)
  Interventions: Drug: Insulin lispro A
- Insulin lispro B (Active Comparator): 20 units (U) subcutaneously (SC)
  Interventions: Drug: Insulin lispro B

INTERVENTIONS:
Drug: Insulin lispro A — 20 units (U) subcutaneously (SC).
  Other Names: LY275585
  Arms: Insulin Lispro A
Drug: Insulin lispro B — 20 U subcutaneously (SC).
  Other Names: LY275585
  Arms: Insulin lispro B

SUMMARY:
This study will compare how the body treats 2 different forms of insulin lispro and how they affect blood sugar levels.

DETAILED DESCRIPTION:
The 2 formulations of insulin lispro will be referred to here as:

Lispro A

Lispro B

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males or females.
* Body mass index (BMI) between 18.5 and 29.9 kilograms per meter squared (kg/m^2)
* Are nonsmokers.
* Have normal blood pressure and pulse rate, a normal electrocardiogram (ECG), and clinical laboratory test results within normal reference range at screening.

Exclusion Criteria:

* History of first-degree relatives known to have diabetes mellitus.
* Evidence of significant active neuropsychiatric disease.
* Evidence of an acute infection with fever or infectious disease.
* Intend to use over-the-counter or prescription medication (apart from vitamin/mineral supplements, occasional paracetamol, or birth control methods).
* Have used systemic glucocorticoids within 3 months prior to entry into the study.
* Have donated blood of 1 unit or more within the last 3 months prior to study entry.
* Excessive alcohol intake
* Have a fasting venous blood glucose (FBG, plasma) >6 millimoles/liter (mmol/L) at screening.
* Have positive hepatitis B surface antigen.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 participants were enrolled into the study. 3 participants discontinued due to subject decision prior to receiving treatment.
Groups:
- Insulin Lispro Dosing Sequence ABAB: Each participant was administered insulin lispro A formulation (Treatment A, test - 2 occasions) and insulin lispro B formulation (Treatment B, reference - 2 occasions) in the dosing sequence ABAB. There was an interval of approximately 4 to 7 days between doses.
- Insulin Lispro Dosing Sequence BABA: Each participant was administered insulin lispro A formulation (Treatment A, test - 2 occasions) and insulin lispro B formulation (Treatment B, reference - 2 occasions) in the dosing sequence BABA. There was an interval of approximately 4 to 7 days between doses.
Period: First Intervention (1 Day )
Arm/Group | Insulin Lispro Dosing Sequence ABAB | Insulin Lispro Dosing Sequence BABA
Started | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0
Period: Interval Between Dosing (4-7 Days)
Arm/Group | Insulin Lispro Dosing Sequence ABAB | Insulin Lispro Dosing Sequence BABA
Started | 20 | 18
Completed | 20 | 17
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention (1 Day)
Arm/Group | Insulin Lispro Dosing Sequence ABAB | Insulin Lispro Dosing Sequence BABA
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0
Period: Interval Between Dosing (4-7 Days)
Arm/Group | Insulin Lispro Dosing Sequence ABAB | Insulin Lispro Dosing Sequence BABA
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Insulin Lispro Dosing Sequence ABAB | Insulin Lispro Dosing Sequence BABA
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0
Period: Interval Between Dosing (4-7 Days)
Arm/Group | Insulin Lispro Dosing Sequence ABAB | Insulin Lispro Dosing Sequence BABA
Started | 20 | 17
Completed | 20 | 16
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Fourth Intervention (1 Day)
Arm/Group | Insulin Lispro Dosing Sequence ABAB | Insulin Lispro Dosing Sequence BABA
Started | 20 | 16
Completed | 20 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Insulin Lispro Dosing Sequence ABAB: Each participant was administered insulin lispro A formulation (Treatment A, test - 2 occasions) and insulin lispro B formulation (Treatment B, reference - 2 occasions) in the dosing sequence ABAB.
- Insulin Lispro Dosing Sequence BABA: Each participant was administered insulin lispro A formulation (Treatment A, test - 2 occasions) and insulin lispro B formulation (Treatment B, reference - 2 occasions) in the dosing sequence BABA.
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro Dosing Sequence ABAB | Insulin Lispro Dosing Sequence BABA | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (7.2) | 34.6 (6.4) | 32.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 20 | 16 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 20 | 18 | 38
  Hispanic or Latino | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter: Area Under the Serum Insulin Concentration Versus Time Curve From Time Zero to the Last Time Point With a Measurable Concentration [AUC0-tlast]
Description: Primary outcome measure is based on the pharmacokinetic area under the concentration-time curve from time 0 to the last time point with a measurable concentration.
Time Frame: 0 up to 8 hours post dose
Population: All participants who had at least one study treatment and had evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole*hour/liter (pmol*h/L)
Groups:
- Insulin Lispro A; Insulin Lispro B: 20 units (U) administered subcutaneously (SC)
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 37 | 38
picomole*hour/liter (pmol*h/L) | 1920 (20) | 1940 (20)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Ratio of geometric least square means = 0.990, 90% CI 2-sided [0.948 to 1.034]

2. Secondary Outcome: Pharmacokinetic Parameter: Maximum Serum Insulin Concentration [Cmax]
Description: The maximum observed insulin lispro concentration following dosing.
Time Frame: 0 to 8 hours post dose
Population: All participants who had at least one study treatment and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole/liter (pmol/L)
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 37 | 38
picomole/liter (pmol/L) | 819 (32) | 887 (34)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Ratio of geometric least square means = 0.933, 90% CI 2-sided [0.897 to 0.972]

3. Secondary Outcome: Pharmacodynamic Parameter: Maximum Glucose Infusion Rate (Rmax)
Description: The maximum observed glucose infusion rate during the euglycemic clamp procedure.
Time Frame: 0 to 8 hours post dose
Population: All participants who had at least one study treatment and had evaluable pharmacodynamic (PD) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per minute (mg/min)
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 37 | 38
milligrams per minute (mg/min) | 544 (23) | 539 (27)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Ratio of geometric least square means = 1.005, 90% CI 2-sided [0.958 to 1.054]

4. Secondary Outcome: Pharmacodynamic Parameter: Time of Maximum Glucose Infusion Rate (tRmax)
Description: Time of maximal glucose infusion rate.
Time Frame: 0 to 8 hours post dose
Population: All participants who had at least one study treatment and had evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 37 | 38
hours | 2.11 (49) | 2.00 (56)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Median Difference (Final Values) = 0.100, 90% CI 2-sided [-0.400 to 0.500]

5. Secondary Outcome: Pharmacodynamic Parameter: Total Amount of Glucose Infused (Gtot)
Description: The total amount of glucose infused during the euglycemic clamp procedure.
Time Frame: 0 to 8 hours post dose
Population: All participants who had at least one study treatment and had evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: grams (g)
Arm/Group | Insulin Lispro A | Insulin Lispro B
Number analyzed (Participants) | 37 | 38
grams (g) | 125 (25) | 123 (30)
Statistical Analysis 1: Comparison: Insulin Lispro A vs Insulin Lispro B; Test type: Superiority or Other; Ratio of geometric least square means = 1.014, 90% CI 2-sided [0.961 to 1.070]

ADVERSE EVENTS:
Description: 38 participants were randomly assigned to treatment, 38 participants received at least 1 dose of study drug, 36 participants completed all 4 periods of the study. One participant only completed 1 insulin lispro B period and then discontinued. This participant did not complete the insulin lispro A periods.
Groups:
- Insulin Lispro A: Insulin lispro A formulation (Treatment A, test - 2 occasions)
- Insulin Lispro B: Insulin lispro B formulation (Treatment B, reference - 2 occasions)
Arm/Group | Insulin Lispro A | Insulin Lispro B
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 9/37 | 12/38
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro A (N=37) | Insulin Lispro B (N=38)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 5 (5) | 4 (6)
Catheter site pain (General disorders) | 1 (1) | 1 (1)
Catheter site swelling (General disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (3) | 1 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes